CLINICAL TRIAL: NCT06497296
Title: The Optimal Timing of the Initiation of Esophagogastroduodenoscopy After Oral Lidocaine Spray
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Hsueh-Chien Chiang, Principal Investigator, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-ER-111-218
Record Dates: First submitted 2024-07-02; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Blood Pressure; Tachycardia
MeSH Terms: conditions — Tachycardia | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Both group accepted 6 puff of lidocaine spray. EGD will be inserted one minute after the lidocaine spray in 1-minute group and 3 minutes waiting in 3-minute group
Who Masked: Participant, Investigator
Masking Description: Sealed and ordered envelope will be opened by assistant and the allocation was written on it. After then, lidocaine spray will be administered. The operator will be informed to prepare 30 seconds before the EGD initiation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-minute group (Placebo Comparator): 6 puff of lidocaine was delivered 1 minute before the initiation of EGD insertion
  Interventions: Drug: Lidocaine
- 3-minute group (Active Comparator): 6 puff of lidocaine was delivered 3 minutes before the initiation of EGD insertion
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Lidocaine spray in both group with same puff number, but the timing before EGD insertion is different

SUMMARY:
Esophagogastroduodenoscopy (EGD) is the main examination in the upper gastrointestinal field. Aspiration pneumonia may happen if choking occurs during the EGD insertion, and the exam quality and efficacy may be affected if gag reflex occurs. The endoscopist may terminate the exam to avoid complications if the patient could not obey the orders. To reach the high quality of EGD examination and to avoid possible complications, the patient's comfort and compliance during the EGD examination are important. Sedation using propofol can improve the patient's comfort and compliance. However, in patients unsuitable for systemic anesthesia, local lidocaine spray at pharynx is performed instead. Until now, there is no standardization of the waiting time between lidocaine spray and the initiation of EGD. This study aimed to investigate the optimal timing of the initiation of esophagogastroduodenoscopy after lidocaine spray.

DETAILED DESCRIPTION:
This study compares the 1-minute waiting time and 3-minute waiting time between the lidocaine spray and the EGD initiation. During the topical anesthesia stage, investigators give local spray with 6 puff on pharynx at the 0 minute in both groups. After the waiting time, EGD is inserted.

The baseline heart rate and blood pressure were recorded before EGD and during the EGD passing through pharynx respectively. After the whole procedure, enrolled patients will fill in the EGD quality questionnaire.

Through this study, investigators can figure out whether 1 minute or 3 minutes may be the optimal waiting time after lidocaine spray.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants included patients aged ≥ 20 years who scheduled EGD from OPD for dyspepsia, peptic ulcer disease, GERD, subepithelial lesion evaluation, and diarrhea

Exclusion Criteria:

* GI bleeding
* endoscopic submucosal dissection due to prolonged scheduled procedure time
* patients from emergency department or ward

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate change | 1 day
  The increase level of heart rate between baseline and during the pharynx insertion of EGD
Blood pressure change | 1 day
  The increase level of systolic blood pressure between baseline and during the pharynx insertion of EGD

SECONDARY OUTCOMES:
EGD comfort quality questionnaire score | 1 day
  comfort quality questionnaire will be written by an assistant and the patient after the EGD procedure. The score includes pain feeling (1-5 points), nausea sensation (1-5 points), abdominal fullness (1-5 points). A higher score indicates more discomfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Hsueh-Chien Chiang, Tainan, Other (Non U.s.), Taiwan

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared after publication
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Result] Rizk MK, Sawhney MS, Cohen J, Pike IM, Adler DG, Dominitz JA, Lieb JG 2nd, Lieberman DA, Park WG, Shaheen NJ, Wani S. Quality indicators common to all GI endoscopic procedures. Gastrointest Endosc. 2015 Jan;81(1):3-16. doi: 10.1016/j.gie.2014.07.055. Epub 2014 Dec 2. No abstract available. PMID 25480102
- [Result] ASGE Standards of Practice Committee; Ben-Menachem T, Decker GA, Early DS, Evans J, Fanelli RD, Fisher DA, Fisher L, Fukami N, Hwang JH, Ikenberry SO, Jain R, Jue TL, Khan KM, Krinsky ML, Malpas PM, Maple JT, Sharaf RN, Dominitz JA, Cash BD. Adverse events of upper GI endoscopy. Gastrointest Endosc. 2012 Oct;76(4):707-18. doi: 10.1016/j.gie.2012.03.252. No abstract available. PMID 22985638
- [Result] Lazzaroni M, Bianchi Porro G. Preparation, premedication, and surveillance. Endoscopy. 2005 Feb;37(2):101-9. doi: 10.1055/s-2004-826149. PMID 15692924
- [Result] Leitch DG, Wicks J, el Beshir OA, Ali SA, Chaudhury BK. Topical anesthesia with 50 mg of lidocaine spray facilitates upper gastrointestinal endoscopy. Gastrointest Endosc. 1993 May-Jun;39(3):384-7. doi: 10.1016/s0016-5107(93)70110-8. PMID 8514070
- [Result] Evans LT, Saberi S, Kim HM, Elta GH, Schoenfeld P. Pharyngeal anesthesia during sedated EGDs: is "the spray" beneficial? A meta-analysis and systematic review. Gastrointest Endosc. 2006 May;63(6):761-6. doi: 10.1016/j.gie.2005.11.059. PMID 16650534
- [Result] Hwang SH, Park CS, Kim BG, Cho JH, Kang JM. Topical anesthetic preparations for rigid and flexible endoscopy: a meta-analysis. Eur Arch Otorhinolaryngol. 2015 Feb;272(2):263-70. doi: 10.1007/s00405-014-3012-8. Epub 2014 Mar 29. PMID 24682602
- [Result] Martin-Marcos I, Fernandez-Morte N, Balsategui-Martin M, Ortiz-Cantero A, Bermudez-Ampudia C, Lopez-Picado A, Perez-Vaquero P, Salvador-Perez M, Cristobal-Dominguez E. Evaluation of pharyngeal lidocaine anesthesia for esophagogastroduodenoscopy: Double-blind randomized control trial. Dig Endosc. 2022 May;34(4):808-815. doi: 10.1111/den.14168. Epub 2021 Nov 17. PMID 34644419
- [Derived] Chiang HC, Chiang CM, Chang WL, Lin MY. Clinical Trial: The Optimal Timing of the Endoscope Insertion After Oral Lidocaine Spray. A Randomized Controlled Trial. J Gastroenterol Hepatol. 2025 Jun;40(6):1428-1434. doi: 10.1111/jgh.16958. Epub 2025 Apr 1. PMID 40166898